CLINICAL TRIAL: NCT06488898
Title: Abdominal Aortic Aneurysm Stabilization With Truncal Cells: Controlled Clinical Trial With Historical Cohorts
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Collaborators: Grupo Dermatologico Y Estetico Pedro Jaen S.A. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HULP-STEM-EVAR-2020
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Aortic Aneurysm, Abdominal
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Phase IIa, single-center clinical trial compared with historical cohorts to evaluate the preliminary safety and efficacy of an allogeneic adipose tissue-derived mesenchymal stem cells infusion in an aneurysmal sac for the treatment of AAA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic adipose tissue-derived mesenchymal stem cells (Experimental): Allogeneic adipose tissue-derived mesenchymal stem cells and expanded, which are considered an "advanced therapy medicinal product" according to European regulation (Regulation (EC) No 1394/2007).
  Interventions: Drug: Allogeneic adipose tissue-derived mesenchymal stem cells

INTERVENTIONS:
Drug: Allogeneic adipose tissue-derived mesenchymal stem cells — Investigational medicinal product: Allogeneic adipose tissue-derived mesenchymal stem cells and expanded, which are considered an "advanced therapy medicinal product" under European regulation (Article 2(1) of Regulation (EC) No 1394/2007 of the European Parliament and the Council of November 13 th 2007 about advanced therapy medicinal products and amending Directive 2001/83/EC and Regulation (EC) No 726/2004).
  Administration form: Local injection by means of a catheter placed inside the previously excluded aneurysmal sac.
  Administration dose: 1x10000000 cells/kg patient weight.
  Administration guidelines: single infusion on the endovascular day AAA intervention.

SUMMARY:
Phase IIa, single-center clinical trial compared with historical cohorts to evaluate the preliminary safety and efficacy of an allogeneic adipose tissue-derived mesenchymal stem cells infusion in an aneurysmal sac for the treatment of AAA.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with AAA greater than 5 cm diameter with endovascular treatment indication, analyzed by aortic AngioCT.
2. Subjects ≥ 18 years at the time of inclusion.
3. Subjects with a good infrarenal neck for a standard device placement, neither fenestrated nor branched.
4. Patients with an estimated life expectancy greater than 2 years at the time of inclusion.
5. Women with childbearing capacity must have a negative pregnancy test at the time of inclusion and must agree to use highly effective contraceptive methods (diaphragms plus spermicide or male condom plus spermicide, oral contraceptive combined with a second method contraceptive implant, injectable contraceptive, permanent intrauterine device, sexual abstinence or partner with vasectomy) during their study participation.
6. The patient must be able to attend all study visits and comply with all study procedures.

Exclusion Criteria:

1. Patients with unresolved neoplasia history or hematologic disease.
2. Patients with uncontrolled arterial hypertension (≥180/110) at the time of inclusion.
3. Patients with severe heart failure (New York Heart Association [NYHA] IV) or ejection fraction <20%.
4. Patients with malignant ventricular arrhythmias
5. Patients with deep vein thrombosis the last three months
6. Patient with active sepsis at the time of inclusion
7. Patients with acute myocardial infarction or stroke in the previous month
8. Any type of medical or psychiatric illness that, in investigator opinion, could be a reason for exclusion from the study.
9. Patient with major surgery or severe craniocerebral trauma in the 3 months prior to inclusion in the study.
10. Administration of any investigational drug at the time of inclusion or in the 3 months prior
11. Infants or pregnant women
12. Transplanted patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation of the study intervention: | 12 months
  The safety of the treatment will be evaluated using the following parameters:
  1. Proportion of procedure-related adverse events occurring throughout the study.
  2. Proportion of adverse events related to allogeneic mesenchymal stem cells infusión derived from adipose tissue occurred throughout the study.
  3. Proportion of patients with major adverse cerebral and cardiovascular events (MACCE) within 12 months after treatment.

SECONDARY OUTCOMES:
Efficacy evaluation of the study intervention. | 6 months
  Change in size of the aneurysm sac by using imaging tests performed during follow-up (CT and echo Doppler). A reduction of the aneurysm sac maximum diameter greater than or equal to 5mm in a period of 6 months is considered significant.

OTHER OUTCOMES:
Stent migration in study intervention group vs historical cohort. | 12 months
  Percentage of patients with stent migration compared to historical cohort.
Presence of leaks on CT control in study intervention group vs historical cohort. | 12 months
  Percentage of patients with presence of leaks on CT control at 1 month and a year compared to historical cohort.
Reoperation at 1 year in study intervention group vs historical cohort. | 12 months
  Reoperation rate at 1 year compared to historical cohort.
Hospital admission in study intervention group vs historical cohort. | 12 months
  Hospital admission rate compared to historical cohort.
Quality of life in study intervention group. | 12 months
  Assessment of change in quality of life: specific quality of life assessment survey at one month and one year after treatment respect to baseline. A 10% change in quality of life scores is considered clinically relevant.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain